CLINICAL TRIAL: NCT05649384
Title: PRospective Evaluation of the European Society of Cardiology 0/1-hour Algorithm's Safety and Efficacy for Triage of Patients With Suspected Myocardial Infarction (PRESC1SE-MI)
Brief Title: Emergency Department Triage of Patients With Acute Chest Pain Based on the ESC 0/1-hour Algorithm (PRESC1SE-MI)
Acronym: PRESC1SE-MI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-02269
Record Dates: First submitted 2022-11-14; First posted 2022-12-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Acute Chest Pain; NSTEMI - Non-ST Segment Elevation MI
Keywords: ESC 0/1-hour algorithm; Emergency department; Chest pain; Chest discomfort; Myocardial Infarction MI; Acute Myocardial Infarction AMI; Acute Coronary Syndrome ACS; NSTEMI Non-ST-segment elevation myocardial infarction; NSTE-ACS Non-ST-segment elevation acute coronary syndrome; Unstable angina; Damaged muscle of the heart; Cardiac Biomarkers; Cardiac Troponin T cTnT; Cardiac-Specific Troponin T; Cardiac Troponin I cTnI; Cardiac-Specific troponin I; Amount of troponin in the bloodstream; Increased troponin level; Elevated troponin level; High troponin level; Troponin assessment; Measurement of troponin levels; High-sensitive troponin test; High-sensitivity troponin T testing; High-sensitive Troponin T hsTnT; cTnT-hs; High-sensitive Troponin I hsTnI; cTnI-hs; High-sensitivity cardiac troponin assays; ED presentation; ED admission; ED work-up; Triage emergency department; Triage emergency room; Triage emergency hospital; Rapid Rule-out of Acute Myocardial Infarction; Shorter stay in the emergency department; ESC 0/3-hour algorithm; ESC Guidelines; European Guidelines; 0/1-hour algorithm; 0/3-hour algorithm
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Emergencies; Chest Pain; Myocardial Infarction; Angina, Unstable | interventions — Algorithms

STUDY DESIGN:
Intervention Model Description: prospective stepped-wedge cluster randomised controlled trial, sites are randomly assigned to either early initiation or late initiation of the ESC hs-cTnT/I 0/1h-algorithm and compared to the standard of care ESC hs-cTnT/I 0/3h-algorith
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0/1-hour algorithm (Experimental): High-sensitivity cardiac troponin (hs-cTn) blood tests are performed at admission (0 h) and 1 hour later in the emergency department.
  Interventions: Diagnostic Test: European Society of Cardiology hs-cTnT/I 0 h/1 h algorithm
- 0/3-hour algorithm (Active Comparator): High-sensitivity cardiac troponin (hs-cTn) blood tests are performed at admission (0 h) and 3 hours later in the emergency department.
  Interventions: Diagnostic Test: European Society of Cardiology hs-cTnT/I 0 h/3 h algorithm

INTERVENTIONS:
Diagnostic Test: European Society of Cardiology hs-cTnT/I 0 h/1 h algorithm — High-sensitivity cardiac troponin (hs-cTn) blood tests are performed at admission (0 h) and 1 hour later in the emergency department.
  Other Names: 0/1-hour algorithm
  Arms: 0/1-hour algorithm
Diagnostic Test: European Society of Cardiology hs-cTnT/I 0 h/3 h algorithm — High-sensitivity cardiac troponin (hs-cTn) blood tests are performed at admission (0 h) and 3 hours later in the emergency department.
  Other Names: 0/3-hour algorithm
  Arms: 0/3-hour algorithm

SUMMARY:
The PRESC1SE-MI study compares two algorithms for triage of patients presenting with chest pain and symptoms of heart attack (myocardial infarction) to the emergency department. Both algorithms are recommended by the European Society of Cardiology: the 0/3-hour algorithm and the 0/1-hour algorithm.

Currently, most emergency departments worldwide use the 0/3-hour troponin algorithm. Cardiac troponin (cTn) is a heart-specific biomarker which indicates damage of the heart muscle and which increases after a heart attack. In the 0/3-hour algorithm, the amount of troponin in the bloodstream is measured with a high-sensitivity assay at admission and 3 hours thereafter. Likewise, the 0/1-hour algorithm means that the blood sample in which the troponin is measured is collected at admission and 1 hour later. Since recent clinical studies suggest that the 0/1-hour algorithm is superior to the 0/3-hour algorithm, many hospitals consider switching to the 0/1-hour algorithm.

The aim of this study is to assess how feasible the time-saving 0/1-hour algorithm would be in reality and whether it provides the same accuracy and safety in the diagnosis of myocardial infarction as the current practice the 0/3-hour algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above
* Presentation with acute non-traumatic acute chest pain to the emergency department
* Suspicion of acute myocardial infarction

Exclusion Criteria:

* Terminal kidney failure requiring dialysis
* Cardiac arrest
* Cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64374 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality or new AMI (type 1) occurring within 30 days of index presentation | 30 days
  Mortality rate and number of newly diagnosed AMI (type 1) in all enrolled patients
Time from ED presentation to ED discharge or transfer | 30 days
  Length of stay in the ED measured in hours

SECONDARY OUTCOMES:
Proportion of patients managed as outpatients | 24 hours
  Number of patients who stay in hospital for index event less than 24 hours
Readmission for suspected AMI within 30 days after index presentation | 30 days
  Number of patients who stay in hospital for a new suspected AMI more than 24 hours within 30 days of index presentation
All-cause mortality at 30 days in all patients | 30 days
  Number of deceased patients within 30 days after index presentation
All-cause mortality at 365 days in all patients | 365 days
  Number of deceased patients within 365 days after index presentation
New AMI (type1) at 30 days in all patients | 30 days
  Number of newly diagnosed AMI (type 1) in all patients within 30 days of index presentation
New AMI (type 1) at 365 days in all patients | 365 days
  Number of newly diagnosed AMI (type 1) in all patients within 365 days of index presentation
Composite of all-cause mortality or new AMI (type 1) at 365 days after index presentation | 365 days
  Mortality rate and number of newly diagnosed AMI (type 1) in all enrolled patients
Satisfaction of patients with their evaluation in the ED | 30 days
  Satisfaction will be measured on a numerical/visual analogue scale from 0-100%, the higher the score, the greater the satisfaction
Treatment costs in the ED | 365 days
  Costs of procedures performed in the ED will be calculated according to national remuneration systems
Length of stay in the ED | 30 days
  Length of stay from admission to the ED to discharge or transfer will be calculated according to national remuneration systems
Feasibility of the 0/1-hour algorithm | 80 minutes
  Feasibility defined as the percentage of patients in whom the "1h" blood draw is performed within 1h +/- 20 minutes from the "0h" blood draw
Effectiveness of rule-in | 30 days
  Effectiveness defined as the time from presentation to coronary angiography in patients ultimately diagnosed with AMI (type 1)
Effectiveness of rule-out | 30 days
  Effectiveness defined as time from presentation to discharge in patients ultimately diagnosed with non-cardiac disease

CONTACTS AND LOCATIONS:
Overall Officials: Christian Müller, MD Prof., Principal Investigator — University Hospital, Basel, Switzerland; Jasper Boeddinghaus, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (20):
- Baylor St. Luke's Medical Center, Houston, Texas, United States
- St Andrew's War Memorial Hospital Brisbane, Brisbane, Australia
- Vienna General Hospital (AKH Wien), Vienna, Austria
- University Central Hospital Helsinki, Helsinki, Finland
- Attikon General Hospital Athens, Athens, Greece
- Italy (3):
  - Careggi University Hospital Florence, Florence
  - Azienda Ospedaliera San Giovanni Addolorata, Roma
  - Hospital Città della Salute e della Scienza di Torino, Torino
- Emergency Institute for Cardiovascular Diseases C.C. Iliescu, Bucharest, Romania
- Konkuk University Medical Center, Seoul, South Korea
- Spain (4):
  - Hospital Clinic Barcelona, Barcelona
  - University Hospital October 12 Madrid, Madrid
  - University Hospital Ramon y Cajal, Madrid
  - Hospital Clínico Universitario Valencia, Valencia
- Switzerland (4):
  - Kantonsspital Aarau, Aarau
  - St. Claraspital, Basel
  - Kantonsspital Luzern, Lucerne
  - University Hospital Zurich, Zurich
- United Kingdom (2):
  - Royal London Hospital, London
  - Royal Cornwall Hospitals Treliske, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boeddinghaus J, Bima P, Crisanti L, Keller DI, Slankamenac K, Christ M, Schuetz P, Wiencierz A, Strebel I, Reinhardt J, Vyshnevska I, Tsao TY, Mahfoud F, Ruggieri MP, Steuer S, Miro O, Harjola VP, Morello F, Nazerian P, Roth D, Zamorano JL, Gannon DE, Pott J, Abubakr MO, Yang HS, Young J, Bicette R, Cuculici A, Bueno H, Sanchis J, Mueller C; PRESC1SE-MI investigators. PRospective evaluation of the European Society of Cardiology 0/1h-algorithm;s safety and efficacy for triage of patients with suspected myocardial infarction (PRESC1SE-MI): Rationale and design of a prospective international multicenter stepped-wedge cluster randomized controlled trial. Am Heart J. 2026 Feb;292:107299. doi: 10.1016/j.ahj.2025.107299. Epub 2025 Oct 31. PMID 41177204